CLINICAL TRIAL: NCT01460420
Title: European Myeloma Network Sequential Phase I / Phase II Trial on RIC Allogeneic Transplantation: an Optimized Program for High Risk Relapsed Patients
Brief Title: Sequential Trial on Reduced Intensity Conditioning (RIC) Allogeneic Transplantation
Acronym: EMN-alloRIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN-alloRIC2010
Record Dates: First submitted 2011-09-22; First posted 2011-10-26 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Hematologic Malignancies; Multiple Myeloma
Keywords: Allogeneic transplantation; Hematologic malignancies; Multiple myeloma; RIC (Reduced Intensity Conditioning)
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + Lenalidomide (Experimental): After conditioning treatment and graft versus host disease prophylaxis with Bz 1.3 mg/m2 on days +1, +4 and +7 plus sirolimus/rapamycin at a dose of 6 mg po on day -5 and then 4 mg per day in order to maintain serum levels in the range of 6-12 ng /mL, a maintenance therapy with Bz 1.3 mg/m2 on days 1, 8 and 15 in cycles of 56 days up to 6 cycles post-transplant and on day +180 Len will be started at a dose of 5 mg and will be maintained until relapse.
  Interventions: Drug: Bz (Bortezomib); Drug: Len (lenalidomide)

INTERVENTIONS:
Drug: Bz (Bortezomib) — Bz 1.3 mg/m2 on days +1, +4 and +7. Maintenance therapy and dose reduction pre-specified.
  Other Names: Codenamed PS-341; Marketed as Velcade
Drug: Len (lenalidomide) — Len at a dose of 6 mg po on day -5 and then 4 mg per day in order to maintain serum levels in the range of 6-12 ng /mL.
  Maintenance therapy and dose reduction pre-specified.
  Other Names: Rapamycin; CC-5013; Marketed as Revlimid

SUMMARY:
The aim of the current study is to improve the outcome of patients with hematologic malignancies (in a phase I trial) and more specifically multiple myeloma (in a phase II trial) by 2 interventions: reduce the risk of graft-versus-host disease (GVHD) and improve the efficacy of the procedure decreasing the risk of relapses after transplant.

Currently, the standard approach used in most centers to prevent graft-versus-host disease after allogeneic transplantation is based on the combination of a calcineurin inhibitor (cyclosporine or tacrolimus) plus a short course of methotrexate. Unfortunately, this strategy is far from ideal, since the risk of acute GVHD is in the range of 30-40% among patients receiving a matched related donor transplantation and even higher among patients receiving transplantation from an unrelated donor while the incidence of chronic GVHD is 60-70% among patients receiving peripheral blood progenitor cells from either a related or unrelated donor.

As far as the patients with multiple myeloma (MM) is concerned, although the development of new drugs has markedly changed the outcome and management of these patients, allogeneic transplantation so far appears to be the only curative option, especially among those patients relapsing after first line treatment. Nevertheless, still new strategies within the allogeneic transplant setting are needed to improve its results.

Relapses may occur either extramedullary (very common in this setting) or systemic. In order to reduce the risk of systemic relapses the investigators will use maintenance therapy with Lenalidomide (Len) which, together with bortezomib (Bz) should contribute to eradicate minimal residual disease (MRD). In case the patient do not obtain complete remission or near complete remission after transplant, in addition to the maintenance therapy, the investigators will use four intensification cycles with VRD (Bz-Len-Dexamethasone).

In summary, the goal is to optimize the efficacy of allogeneic transplantation by two interventions: one focused on reducing the risk of relapse and the other on reducing the incidence of GVHD.

ELIGIBILITY:
Inclusion Criteria:

Phase I: For the first 10 patients:

* Patients with any haematological malignancy in > CR1 (first complete remission)
* Suitable related donor human leukocyte antigen (HLA)identical
* Age > 18 and < 70 years

For the 10 subsequent patients:

* Patients with any haematological malignancy candidates to receive an allogeneic transplant
* Suitable related or unrelated donor (a maximum of 1 mismatched is allowed)
* Age > 18 and < 70 years phase II trial:
* High-risk multiple myeloma patients at first relapse / second complete remission candidates to receive an allogeneic transplantation
* Age:> 18 < 70 years.
* Suitable donor, related or unrelated (a maximum of 1 mismatched is allowed)
* Measurable disease
* High risk first relapse is defined as:
* First early relapse after Autologous Stem Cell Transplant (ASCT)< 24 months
* First late relapses in case the patient does not achieve CR after second ASCT
* First relapse in patients with poor cytogenetic features
* All subjects must be able to comply with the Lenalidomide Pregnancy Prevention Risk Management Plan.

Exclusion Criteria:

Any of the following:

* Prior severe comorbidity such as:

  * Heart failure or previous infarction
  * Uncontrolled Hypertension
  * Arrhythmia
  * Cirrhosis
* Peripheral neuropathy >Grade 2, 14 days prior to inclusion
* Psychiatric disease
* Prior history of other neoplasia except for carcinoma in situ in the last 10 years
* Hypersensitivity to Bz, Boric acid mannitol.
* Patients unable to use appropriate contraceptive methods
* Patients who have received an investigational drug 30 days prior to inclusion
* Positive human immunodeficiency virus (HIV) or active viral hepatitis
* Patients with pericardial disease
* Patients with acute diffuse infiltrative pulmonary disease
* Patients not willing to comply with the Lenalidomide Pregnancy Prevention Risk Management Plan
* Patients not willing to receive thromboprophylaxis during the consolidation phase will not be eligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Phase I trial: Safety of Len + Bz in patients with hematologic malignancies Phase II trial: Safety and efficacy of an optimized strategy of allogeneic transplantation in multiple myeloma undergoing allogeneic transplantation. | Up to one year after transplant
  For phase I trial: safety of Len + Bz. The phase I trial safety criteria will be evaluated in terms of (1) engraftment defined as > 500 granulocytes / microL and > 20.000 platelets / microL x 3 consecutive days will be required for 9/10 patients, (2) incidence of neuropathy grades 3-4 attributed to Bz > 20% (3) incidence of gastrointestinal toxicity attributed to Bz > 20%.
  For phase II trial: safety evaluated through adverse events and toxicity and efficacy evaluated as reduction of relapse rate as defined by the EBMT criteria.

SECONDARY OUTCOMES:
Incidence of GVHD with this combination (phase I and II) | Up to one year after transplant
  Evaluation of a novel combination of Bz plus Len to prevent GVHD after allogeneic transplantation in patients with haematologic malignancies/MM
Phase II: response and relapse rate of this approach | Up to one year after transplant
  Reduction of relapse rate as defined by the EBMT (European Group for Blood, and Marrow Transplant)criteria.
Phase II: safety of the procedure | Up to one year after transplant
  For all patients safety will be assessed by the reporting of adverse events starting with the first study-related procedure and up to 30 days after the treatment period. The severity of adverse events will be assessed using National Cancer Institute (NCI) common toxicity criteria (CTC).
Evaluate the efficacy on survival | Up to one year after transplant
  Evaluate the efficacy of the procedure in terms of event free and overall survival
Efficacy of positron emission tomography (PET scan)and local radiotherapy | Up to one year after transplant
  Analyze the prognostic value and efficacy of imaging studies using PET scan and local radiotherapy in involved fields prior to or after (> 100 days) conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Antonio Perez-Simon, MD-PhD, Principal Investigator — University Hospital Virgen del Rocio
Locations (10):
- Medizinische Klinik and Poliklinik II, University Hospital, Würzburg, Germany
- Italy (2):
  - S Giovanni Battista Hospital, Torino
  - Azienda Ospedaliera Universitaria di Udine, Udine
- Spain (6):
  - Hospital Clinic i Provincial,, Barcelona
  - Hospital Santa Creu I Sant Pau,, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Gregorio Marañón,, Madrid
  - Hospital Clinico Universitario Salamanca,, Salamanca
  - Hospital Universitario Virgen del Rocío,, Seville
- Karolinska University Hospital, Huddinge, Stockholm, Sweden